CLINICAL TRIAL: NCT01645878
Title: Effect of Education on Breast Feeding on Primiparous Women
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sedigeh Azhari, Faculty member, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Hands on and hands off
Record Dates: First submitted 2012-07-17; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2010-01

CONDITIONS: Breastfeeding
Keywords: Primiparous Mothers; self-efficacy,; hands off,; hands on ,; social cognitive theory
MeSH Terms: conditions — Breast Feeding | interventions — Therapeutic Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hands on (Experimental): breast feeding instructed by direct help of instructor
  Interventions: Behavioral: hands on
- hands off (Experimental)
  Interventions: Behavioral: hands off
- Control (Other): Routin breast feeding education
  Interventions: Behavioral: routin breast feeding education

INTERVENTIONS:
Behavioral: hands on — in hands on group it was instructed by direct help of instructor, mothers could ask questions and if necessary it was done again by researcher.
  Arms: Hands on
Behavioral: hands off — In hands off group, was instructed by pictures, if mothers had questions, they could watch the pictures again
  Arms: hands off
Behavioral: routin breast feeding education
  Arms: Control

SUMMARY:
Exclusive breastfeeding is very important for an infant's growth and development. Self-efficacy is a modifiable psychological variable in sustained breastfeeding that is defined as a mother's confidence in her perceived ability about successful exclusive breastfeeding. Self- efficacy beliefs function as an important set of human motivation , affect , and action which operate on action, through motivation, cognitive and affective interventing process. teaching strategies ,based on Bandura,s self-efficacy theory and adult learning principles were incorporated in this research design. In regards with the importance of education in increasing breastfeeding self-efficacy and exclusive breastfeeding, the current study was conducted in order to compare of the effectiveness of two educational methods, i.e., "Hands on" and" Hands off" on breastfeeding self-efficacy in primiparous mothers.

In the present clinical trial, 136 nursing mother were randomly assigned to one of the three groups. Participants in the experimental groups received one of the structured one-on-one educational sessions (i.e., hands off or hands on) within the first two hours of giving birth. Mothers in control group received usual postpartum care. Follow-up assessments were conducted one, four, and eight weeks after the birth. Data collection was done through interview forms, examination and observation, checklist of breastfeeding status, breastfeeding self-efficacy and daily-feeding form.

ELIGIBILITY:
Inclusion Criteria:

vaginal normal delivery normal neonate lack of maternal- neonatal lactation problems contact number satisfying in participation in study

Exclusion criteria would not like to continue used tranquilizers or experienced stressful events

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Breast feeding self-efficacy | up to 2 month